CLINICAL TRIAL: NCT05718700
Title: A Registry Study of Treatment With Bulevirtide in Participants With Chronic Hepatitis D Infection
Brief Title: Study of Bulevirtide in Participants With Chronic Hepatitis D Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-589-6206; 2022-501901-10 (Other: European Medicines Agency)
Expanded Access: NCT06780579 (Available)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis D Infection
MeSH Terms: interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 144 Weeks
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bulevirtide (previously participated in Study MYR-Reg-2): Participants who are currently receiving bulevirtide (BLV) according to the approved label and have participated in Study MYR-Reg-02.
  Interventions: Drug: Bulevirtide
- Bulevirtide: Participants who are scheduled to receive BLV according to the approved label.
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — Administered via subcutaneous (SC) injections
  Other Names: Hepcludex®

SUMMARY:
The main goal of this study is to collect post marketing data from patients with chronic hepatitis D virus (HDV) infection who are treated with bulevirtide to describe the long-term effects of bulevirtide treatment and evaluate the safety of participants treated with bulevirtide.

DETAILED DESCRIPTION:
The study design time perspective is retrospective and prospective for participants who previously participated in MYR-Reg-02 and are currently receiving BLV and prospective for participants who are scheduled to receive BLV.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals who have been diagnosed with chronic hepatitis D virus (HDV) infection for at least 6 months before study enrollment, confirmed by respective documentation in the individuals' medical records.
* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Must be willing and able to comply with the visit schedule and study requirements.
* Cohort 1 only: Must have participated in study MYR-Reg-02.
* Cohort 2 only: Individuals scheduled to receive bulevirtide (BLV) according to the approved label or for whom the decision to start treatment with BLV according to the approved label has been made and treatment initiation is planned.

Key Exclusion Criteria:

* Individuals currently enrolled in BLV clinical treatment studies and/or other interventional clinical studies with an investigational agent.
* History or current presence of clinically significant illness or any other major medical disorder that may interfere with individual follow-up, assessments, or compliance with the protocol.
* Coinfection with hepatitis C virus (HCV) or human immunodeficiency virus (HIV) (Individuals with HCV antibodies can be enrolled if HCV RNA is negative).
* Solid organ transplantation.
* Any history, or current evidence of clinical hepatic decompensation (ie, ascites, encephalopathy, jaundice, or gastrointestinal bleeding (GIB)).
* Presence of hepatocellular carcinoma (HCC) as evidenced by imaging (eg, ultrasound or computed tomography scan) performed within 4 months prior to Day 1 for individuals with cirrhosis and within 6 months prior to Day 1 for individuals without cirrhosis.
* Pregnant or breastfeeding females.
* Individuals with a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed by a positive polymerase chain reaction test result.
* Known hypersensitivity or contraindication to BLV or formulation excipients.
* Individuals who are committed to an institution by virtue of a court or official order.
* Individuals deemed by the study investigator to be inappropriate for study participation for any reason not otherwise listed. This includes persons dependent on the sponsor, investigator, or trial site.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants who participated in Study MYR-Reg-02 or are scheduled to receive BLV according to the approved product label and not currently enrolled in a clinical treatment study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Exposure-adjusted Incidence of Participants With Liver-related Event: Hepatic Decompensation, Hepatocellular Carcinoma (HCC), Liver Transplantation, and Liver-related Death | Up to 144 weeks

SECONDARY OUTCOMES:
Percentage of Participants Who Develop Cirrhosis During The Study Among Participants Who Were Previously Noncirrhotic | Up to 144 weeks
Percentage of Participants With Serious Adverse Events | First dose date up to 144 weeks plus 30 days
Percentage of Participants With Grade 3 or 4 Adverse Events (AEs) | First dose date up to 144 weeks plus 30 days
Percentage of Participants With Discontinuations Due to AEs | First dose date up to 144 weeks plus 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (52):
- Austria (4):
  - Medizinische Universität Graz Universitätsklinik für Innere Medizin, Klinische Abteilung für Gastroenterologie und Hepatologie, Graz
  - Aö Landeskrankenhaus Hall, Hall in Tirol
  - Universitätsklinik für Innere Medizin I Innsbruck, Innsbruck
  - Medizinische Universitat Wien, Vienna
- France (16):
  - Centre Hospitalier Universitaire D'Angers, Angers
  - Hôpital Avicenne - APHP, Bobigny
  - Hopital Beaujon, Clichy
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier Universitaire De Lille- Hôpital Huriez, Lille
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Saint Eloit, Montpellier
  - APHP Hôpital Pitié Salpêtrière, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier De Perigueux, Périgueux
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital Charles-Nicolle - CHU de Rouen, Rouen
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
- Germany (12):
  - Leber- und Studienzentrum Checkpoint, Berlin
  - Charité. Univeritätsmedizin Berlin, CMM & CVK, Department of Hepatology and Gastroenterology, Berlin
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I, Bonn
  - Universitätsklinikum Düsseldorf, Klinik für Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Universitätsklinikum Gießen und Marburg - Gießen, Medizinisch Klinik V, Giessen
  - IFI- Institut für interdisziplinäre Medizin, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Liver Study Centre Kiel, Kiel
  - Klinikum rechts der Isar der Technischen Universität München, Munich
  - St Josephs-Hospital Wiesbaden, Med Klinik 2, Wiesbaden
- Romania (10):
  - Dr. Victor Babes Clinical Hospital for Infectious and Tropical Diseases, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Prof. Dr. Agrippa Ionescu Emergency Clinical Hospital, Bucharest
  - National Institute of Infectious Diseases "Prof. Dr. Matei Balş", Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova
  - GastroMedica SRL, Iași
  - Hospital for Infectious Diseases St. Cuvioasa Paraschiva, Iași
  - Clinical Hospital for Infectious Diseases and Pneumophthisiology Dr. Victor Babe, Timișoara
  - Emergency County Clinical Hospital "Pius Brînzeu" Timişoara, Timișoara
- Spain (7):
  - Complejo Hospitalario Torrecárdena, Almería
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario La Paz. Paseo de la Castellana 261, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-589-6206